CLINICAL TRIAL: NCT01811498
Title: Phase I/II Trial of Repeated Super-Selective Intraarterial Cerebral Infusion of Bevacizumab (Avastin) for Treatment of Newly Diagnosed Glioblastoma Multiforme
Brief Title: Repeated Super-Selective Intraarterial Cerebral Infusion of Bevacizumab (Avastin) for Treatment of Newly Diagnosed GBM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Feinstein Institute for Medical Research (Other)
Responsible Party: Principal Investigator, John Boockvar, MD Zucker SOM @Hofstra/Northwell, Professor, Feinstein Institute for Medical Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-352
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Glioblastoma Multiforme; Brain Tumor
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SIACI of Bevacizumab (Experimental): Superselective Intraarterial Cerebral Infusion (SIACI) of Bevacizumab
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab
  Other Names: Avastin

SUMMARY:
The high-grade malignant brain tumors, glioblastoma multiforme (GBM), comprise the majority of all primary brain tumors in adults. This group of tumors also exhibits the most aggressive behavior, resulting in median overall survival of only 9-12 months. Initial therapy consists of either surgical resection, external beam radiation, or both. All patients experience a recurrence after first-line therapy, so improvements in both first-line and salvage therapy are critical to enhancing quality-of-life and prolonging survival. It is unknown if currently used intravenous (IV) therapies even cross the blood brain barrier (BBB). We have shown in a previous phase I trial that a single Superselective Intraarterial Cerebral Infusion (SIACI) of Bevacizumab (up to 15mg/kg) is safe and effective in the treatment of recurrent GBM. Therefore, this phase I/II clinical research trial is an extension of that trial in that we seek to test the hypothesis that repeated dosing of intra-arterial Bevacizumab is safe and effective in the treatment of newly diagnosed malignant glioma. By achieving the aims of this study we will also determine if repeated intra-arterial Bevacizumab improves progression free and overall survival in newly diagnosed patients. We expect that this project will provide important information regarding the utility of repeated SIACI Bevacizumab therapy for malignant glioma, and may alter the way these drugs are delivered to our patients in the near future.

DETAILED DESCRIPTION:
The experimental aspects of this experimental plan will include:

1. Subjects will first be treated with Mannitol prior to chemotherapy infusion (Mannitol 20%; delivered IA, 12.5 mL over 2 minutes) in order to disrupt the blood brain barrier. This technique has been used in several thousand subjects in previous studies for the IA delivery of chemotherapy for malignant glioma.
2. Subjects will then be treated with repeated intraarterial delivery (SIACI) of Bevacizumab. Each subject will receive one dose of IA Bevacizumab on day 30, followed by chemoradiation. SIACI of Bevacizumab will be repeated every three months for a total of 3 infusions.

ELIGIBILITY:
Criteria for Inclusion:

* Male or female patients of ≥18 years of age.
* Patients with documented histologic diagnosis of glioblastoma multiforme (newly diagnosed)
* Patients must have at least one confirmed and evaluable tumor site.∗

  *A confirmed tumor site is one which is biopsy-proven. NOTE: Radiographic procedures (e.g., Gd-enhanced MRI or CT scans) documenting existing lesions must have been performed within three weeks of treatment on this research study.
* Patients must have a Karnofsky performance status ≥70% (or the equivalent ECOG level of 0-2) and an expected survival of ≥ three months.
* Patients must agree to use a medically effective method of contraception during and for a period of three months after the treatment period. A pregnancy test will be performed on each premenopausal female of childbearing potential immediately prior to entry into the research study.

Criteria for Exclusion:

* Previous treatment with Bevacizumab.
* Women who are pregnant or lactating.
* Women of childbearing potential and fertile men who decline to use effective contraception during and for a period of three months after the treatment period.
* Patients with significant intercurrent medical or psychiatric conditions that would place them at increased risk or affect their ability to receive or comply with treatment or post-treatment clinical monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2021-08 (Actual); Study Completion 2021-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Boockvar, MD, Principal Investigator — Feinstein Institute for Medical Research
Locations (1):
- Lenox Hill Brain Tumor Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SIACI of Bevacizumab: Superselective Intraarterial Cerebral Infusion (SIACI) of Bevacizumab
  Bevacizumab
Period: Overall Study
Arm/Group | SIACI of Bevacizumab
Started | 31
Completed | 23
Not Completed | 8

BASELINE CHARACTERISTICS:
Population: A total of 31 patients with newly diagnosed GBM were screened and enrolled in the trial between February 2013 and Dec 2019. As the trial was designed to test the safety and efficacy of repeated dosing, only those patients receiving 2 or 3 IA treatments with BV in addition to standard therapy were considered evaluable. Twenty-three patients with newly diagnosed GBM were included in the final analysis.
Arm/Group | SIACI of Bevacizumab
Number analyzed (Participants) | 23
Age, Continuous [Median (Standard Deviation); unit: years] | 65 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 17
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined from the date of the first dose of SIACI Bevacizumab until first documentation of disease pro- gression, or death from any cause, whichever occurred first.
Time Frame: Percent of Participants with 6 Month Progression-Free Survival
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SIACI of Bevacizumab
Number analyzed (Participants) | 23
percentage of participants | 91.3 [69.5 to 97.8]

2. Primary Outcome: Overall Survival (OS)
Description: Overall Survival was defined from the date of the first dose of SIACI Bevacizumab until death from any cause.
Time Frame: 8 months, and until death of any cause, up to approximately 8 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SIACI of Bevacizumab
Number analyzed (Participants) | 23
months | 23.1 [12.2 to 36.9]

3. Secondary Outcome: Number of Adverse Events
Description: The descriptive frequency of subjects experiencing toxicities will be tabulated.
Time Frame: 30 days post treatment
Population: Total of 23 participants some who had multiple AE's therefore the adverse events number exceeds particpants.
Measure: Number; unit: Adverse events
Arm/Group | SIACI of Bevacizumab
Number analyzed (Participants) | 23
Adverse events
  Grade 1 Adverse Events | 31
  Grade 2 Adverse Events | 15
  Grade 3 Adverse Events | 12

ADVERSE EVENTS:
Time Frame: Adverse events were assessed up to 30 days post treatment (approximately 8 months). All-Cause Mortality was from first dose until death, approximately 8 years.
Arm/Group | SIACI of Bevacizumab
All-Cause Mortality (participants affected / at risk) | 16/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 16/23
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SIACI of Bevacizumab (N=23)
Fatigue (General disorders) | 7 (7)
Anxiety (General disorders) | 2 (2)
Headache (General disorders) | 2 (2)
Brain Hemorrhage (Nervous system disorders) | 2 (2)
Unilateral Weakness (Nervous system disorders) | 4 (4)
Aphasia (Nervous system disorders) | 6 (6)
Seizure (Nervous system disorders) | 7 (7)
Paresthesia (Nervous system disorders) | 1 (1)
Memory Impairment (Nervous system disorders) | 1 (1)
Appetite Loss (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Gastric Reflux (Gastrointestinal disorders) | 1 (1)
Vasospasm (Vascular disorders) | 1 (1)
Thrombocytopenia (Vascular disorders) | 3 (3)
Deep Vein Thrombosis (Vascular disorders) | 3 (3)
Pulmonary Embolus (Vascular disorders) | 2 (2)
Leukopenia (Vascular disorders) | 1 (1)
Scalp Tenderness (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Creatinine Increase (Metabolism and nutrition disorders) | 1 (1)
GGT Increase (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT01811498/Prot_SAP_000.pdf